CLINICAL TRIAL: NCT01693705
Title: Outcome Evaluation of Patients After Percutaneous Tracheostomy Due to Respiratory Failure in an Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0053-12-HYMC
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Respiratory Insufficiency
Keywords: Tracheostomy
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tracheostomy Patients: Critical care patients with respiratory failure who were mechanically ventilated and who underwent tracheostomy
  Interventions: Procedure: Tracheostomy
- Non-Tracheostomy Patients: Critical care patients with respiratory failure who were mechanically ventilated but did not undergo tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy
  Groups: Tracheostomy Patients

SUMMARY:
To determine the morbidity and mortality of patients who have undergone percutaneous tracheostomy due to respiratory failure in the critical care unit and after intensive care in the internal medicine department, including follow-up of quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated critical care patients

Exclusion Criteria:

* All others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure who were mechanically ventilated in the critical care unit
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with tracheostomy due to respiratory failure who died | Six months
  Retrospective review of charts showing increase in morbidity in patients with respiratory failure with tracheostomy taking place 2 weeks after admission to critical care

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel